CLINICAL TRIAL: NCT05360537
Title: Effects of Degludec/Liraglutide on Time in Range, Markers of Inflammation and Endothelial Dysfunction Compared to Scheme Insulin Basal Bolus, in a Population of Diabetic Inpatients and Possible Correlation With Intra-hospital Mortality Rates
Brief Title: Effects of Degludec/Liraglutide on Time in Range, Inflammation and Endothelial Function vs Insulin Basal Bolus in Diabetic Inpatients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Antonino Tuttolomondo, University professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U Palermo
Record Dates: First submitted 2022-04-20; First posted 2022-05-04 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Insulin Degludec/Liraglutide
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec; IDegLira; Insulin Glargine

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider
Masking Description: Double (Participant, Care Provider)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients treated with Insulin Degludec/Liraglutide (Experimental): Diabetes therapy with Insulin Degludec/Liraglutide and various combinations of metformin, repaglinide, sulfonylureas.
  Interventions: Drug: Insulin Degludec / Liraglutide Injectable Product
- patients treated with Insulin regime Basal Bolus (Active Comparator): Diabetes therapy with the combination of a single administration of glargine insulin and three administration of Aspart Insulin.
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: Insulin Degludec / Liraglutide Injectable Product — administration of Insulin Degludec/Liraglutide
  Other Names: Insulin Degludec/Liraglutide
  Arms: patients treated with Insulin Degludec/Liraglutide
Drug: Insulin Glargine — Administration of glargine insulin
  Other Names: glargine
  Arms: patients treated with Insulin regime Basal Bolus

SUMMARY:
The study aims to evaluate the effects of Insulin Degludec/Liraglutide on glycemic variability assessed by continuous glycemic monitoring with the function time in range, serum markers of inflammation, markers of endothelial dysfunction and a possible correlation with intra and extra-hospital mortality rates in a group of hospitalized diabetic patients compared to a control group of in-patient diabetic in treatment on insulin Basal-bolus.

DETAILED DESCRIPTION:
100 patients with type 2 diabetes mellitus were recruited at the Internal Medicine with Stroke care ward of the University hospital of Palermo "P. Giaccone" from April 2022 to April 2024. 50 patients were treated with Insulin Degludec/Liraglutide, 50 were undertaken treatment regime with Insulin Basal Bolus (control group).

The study was carried out in accordance with the principles of the Helsinki Declaration revised in 2001 and all patients gave their written consent to take part in this research.

Each patient treated was compared for age, sex and cardiovascular risk with control patients. The diagnosis of type 2 diabetes mellitus was based on the revised criteria of the American Diabetes Association (ADA), and using a clinical algorithm that considered the age of onset of the disease, the symptoms and weight present, the family history and the therapy practiced. Arterial hypertension was defined according to the 2017 ESC-ESH criteria. Dyslipidemia was defined based on total cholesterol levels> 200 mg/dl, triglycerides> 150 mg/dl and HDL levels <40 mg/dl regardless of the patient's gender.

Among the cases enrolled, 135 (100%) had type 2 diabetes mellitus, 110 (80 %) had arterial hypertension and 74 (55%) hypercholesterolemia.

Clinical and anthropometric data were collected at the time of recruitment. Blood samples were taken from each patient (cases and controls) to determine serum glucose, HbA1c, CRP, Ferritin, IL-6. These withdrawals were then repeated three months and six months from the time of recruitment.

The glycemic variability was assessed by continuous glycemic monitoring with the analysis of Time in Range

The digital endothelial function was evaluated through the RHI-pat analysis using Endo-PAT2000.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type 2
* Mild-moderate Hyperglycemia (180-400 mg/dl)
* Acute events (Pneumonia, Acute cardiac Ischemia, Ictus, IVU)

Exclusion Criteria:

* Diabetes mellitus type 1
* Diabetic ketoacidosis
* Hyperosmolar coma
* Severe hypoglycaemia
* Acute Pancreatitis
* Cancer
* use of corticosteroids
* pregnancy
* Chronic kidney disease (< 30 ml/min) or hemodialysis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Change of Time in Range % at 7 days, at 1 and 6 months | 7 days, 1 months and 6 months
  Evaluation of Time in Range % by continuous glycemic monitoring
Change of hypoglycemic events | 7 days, 1 months and 6 months
  Change of hypoglycemic events (symptoms and serum glycemia < 60 mg/dl)
Change from Baseline Reactive Hyperemia Index at 3 and 9 months | 7 days, 1 months and 6 months
  Change of Endothelial function by the use of Endopat2000 with the evaluation of Reactive Hypereremia Index (normal value of RHI > 1,27)

SECONDARY OUTCOMES:
Change from Baseline serum of C- Reactive-Protein (CRP) | 7 days, 1 months and 6 months
  Variation from baseline serum levels of C- Reactive-Protein (CRP) (mg/dl)
Change from Baseline serum levels of Interleukin-6 (IL6) | 7 days, 1 months and 6 months
  Variation from baseline serum levels of Interleukin-6 (IL6) (pg/ml)
Change from Baseline serum levels of ferritin | 7 days, 1 months and 6 months
  Variation from baseline serum levels of ferritin (mcg/L)
Change of intra and extra-hospital mortality | 7 days, 1 months and 6 months
  Change of intra and extra-hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Tuttolomondo, Professor, Study Director — University of Palermo
Locations (1):
- Internal Medicine Ward, University of Palermo, Palermo, Italy